CLINICAL TRIAL: NCT06772454
Title: To Evaluate the Efficacy and Safety of Inhaled Corticosteroids Combined With Bronchodilators and Programmed Death-ligand 1 (PD-L1) Inhibitor Plus Platinum-based Chemotherapy in Patients With Advanced Lung Squamous Cell Carcinoma Complicated With Chronic Obstructive Pulmonary Disease (COPD)
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Guangzhou Institute of Respiratory Disease
Other Study IDs: CROC202315
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer Squamous Cell; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Antitumor therapy: All patients received suglizumab + paclitaxel + carboplatin: Suglizumab 1200 mg IV Q3W Paclitaxel (albumin-bound) 100 mg/m2 IV, D1, 8, 15, Q3W Carboplatin AUC=5 mg/mL/min IV Q3W A total of 4 administration cycles were given, and Suglizumab 1200 mg IV Q3W was maintained after 4 administration cycles.
  Interventions: Drug: Antitumor therapy
- Inhaled preparation for COPD: 60 patients were randomly assigned to the following two groups in a 1:1 ratio, with about 30 patients in each group. Group A: Receiving a long-acting beta-2 agonist (LABA) + a long-acting anticholinergic (LAMA) combination: Glonium bromide formoterol inhalation aerosol (7.2ug/5ug, trade name: Biwapin, Astrazeneca), 2 inhalations twice a day. Group B: Received inhaled glucocorticoid (ICS) +LABA+LAMA as a three-drug combination: budesonide/glononium bromide/formoterol :160ug/7.2ug/4.8ug, Astrazeneca), 2 inhalations twice daily.
  Interventions: Drug: Inhaled preparation for COPD

INTERVENTIONS:
Drug: Antitumor therapy — All patients received suglizumab + paclitaxel + carboplatin:
  Suglizumab 1200 mg IV Q3W Paclitaxel (albumin-bound) 100 mg/m2 IV, D1, 8, 15, Q3W Carboplatin AUC=5 mg/mL/min IV Q3W A total of 4 administration cycles were given, and Suglizumab 1200 mg IV Q3W was maintained after 4 administration cycles
  Groups: Antitumor therapy
Drug: Inhaled preparation for COPD — 60 patients were randomly assigned to the following two groups in a 1:1 ratio, with about 30 patients in each group.
  Group A: Receiving a long-acting beta-2 agonist (LABA) + a long-acting anticholinergic (LAMA) combination: Glonium bromide formoterol inhalation aerosol (7.2ug/5ug, trade name: Biwapin, Astrazeneca), 2 inhalations twice a day.
  Group B: Received inhaled glucocorticoid (ICS) +LABA+LAMA as a three-drug combination: budesonide/glononium bromide/formoterol :160ug/7.2ug/4.8ug, Astrazeneca), 2 inhalations twice daily.
  Groups: Inhaled preparation for COPD

SUMMARY:
To evaluate the efficacy and safety of inhaled corticosteroids combined with bronchodilators and programmed death-ligand 1 (PD-L1) inhibitor plus platinum-based chemotherapy in patients with advanced lung squamous cell carcinoma complicated with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* This project is a multi-center, randomized controlled, intentionality analysis study.

Inclusion criteria:

1. Age ≥18 years old;
2. Histological or cytological examination confirmed clinically primary squamous non-small cell lung cancer stage IIIB-IV (according to AJCC 8th Edition);
3. Patients with stable moderate to severe chronic obstructive pulmonary disease (COPD) were diagnosed according to the GOLD2021 standard and the Guidelines for Diagnosis and Treatment of Chronic Obstructive Pulmonary Disease (Revised 2021), with blood eosinophils ≤300 /ul and ≥100 /ul;
4. The gene test showed that the driver gene (EGFR/ALK/BRAF/ROS1/KRAS/ HER2/MET/RET /NTRK) was negative;
5. ECOG PS 0-2 points;
6. Clinical evaluation is suitable for suglizumab combined with paclitaxel (albumin-bound) and carboplatin anti-tumor first-line therapy, as well as chronic obstructive pulmonary maintenance therapy with long-acting bronchodilators or inhaled corticosteroids;
7. Clinical records of suglizumab treatment, chemotherapy and other treatments are available;
8. Patients who have previously used bronchodilators and inhaled corticosteroids should undergo a washout period of at least 15 days;
9. Patients voluntarily join the project and sign informed consent;

Exclusion Criteria:

* 10. Concurrent with any malignant active tumor other than squamous non-small cell lung cancer; 11. Prior systematic treatment for advanced/metastatic non-small cell lung cancer; 12. Patients with diseases requiring long-term oral or intravenous use of glucocorticoids, such as autoimmune diseases, asthma, nephritis, type 1 diabetes, hyperthyroidism, etc.; Etc.; 13. Oral or intravenous use of glucocorticoids for any reason within 1 month prior to screening; 14. The patient was assessed by the researchers as having severe liver and kidney dysfunction; 15. Accompanied by acute type I/II respiratory failure or long-term use of non-invasive or invasive ventilator assisted ventilation or frequent acute exacerbations (≥2 times/year of moderate and severe acute exacerbations); 16. Women who are pregnant or nursing, or who are planning to become pregnant; Currently receiving or planning to participate in any other clinical studies;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years, diagnosed with stage IIIb-Ⅳ primary squamous non-small cell lung cancer, diagnosed as stable moderate to severe chronic obstructive pulmonary disease (COPD), genetic testing showed negative driver genes, ECOG PS 0-2 scores, and prior bronchodilators and inhaled corticosteroids were required to undergo a eluting period of at least 15 days. Patients volunteered to join the program.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
PSF、Time and severity of the first acute exacerbation of severe COPD (AECOPD) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- NO.28 Qiaozhong Zhong Road, Liwan District, Guangzhou City, Guangdong Province, Guangzhou, Guangdong, China